CLINICAL TRIAL: NCT00395967
Title: Effect of AMD3100 (240µg/kg) on the Apheresis Yield of CD34+ Cells When Given To Multiple Myeloma or Non-Hodgkin's Lymphoma Patients Predicted to be Unable to Mobilize ≥2 x 10^6 CD34+ Cells in Three Apheresis Days When Given G-CSF Alone
Brief Title: AMD3100 (Plerixafor) in Multiple Myeloma (MM) or Non-Hodgkin's Lymphoma (NHL) Patients Predicted to be Unable to Mobilize With G-CSF Alone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment terminated in 2005 to focus on Phase 3 study enrollment.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-2109
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-08-13 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma; Lymphoma, Non-Hodgkin's
Keywords: Non-Hodgkin's Lymphoma; Multiple Myeloma; stem cell mobilization; autologous transplantation; AMD3100
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Experimental): Patients who were predicted to be unable to mobilize a minimum number of cells (≥2*10^6 CD34+ cells/kg) in 3 apheresis days when given granulocyte colony-stimulating factor (G-CSF) alone and who were eligible for autologous peripheral blood stem cell transplantation.
  Interventions: Drug: G-CSF plus plerixafor

INTERVENTIONS:
Drug: G-CSF plus plerixafor — Mobilization with Granulocyte Colony Stimulating Factor (G-CSF) (10 µg/kg once a day) for 5 days. Patients received once daily plerixafor treatment (240 mg/kg) in the evening (10 to 11 hours prior to apheresis) for up to 3 days if peripheral blood CD34+ cell counts on Day 5 met the entry criteria. Morning doses of G-CSF (10 µg/kg) continued throughout apheresis.
  Other Names: Mozobil; AMD3100

SUMMARY:
This Phase 2 study was designed to assess the safety and hematological activity of AMD3100 (plerixafor) in patients with non-Hodgkin's lymphoma (NHL) or multiple myeloma (MM) who were predicted to be unable to mobilize ≥2*10^6 CD34+ cells/kg within 3 apheresis days. Patients with NHL and MM were eligible to enter the study if they had undergone cyto-reductive chemotherapy, were to undergo autologous transplantation, and met the inclusion/exclusion criteria.

The purpose of this protocol was to determine whether plerixafor in combination with Granulocyte Colony Stimulating Factor (G-CSF) can increase the circulating levels of peripheral blood stem cells (PBSCs) in patients whose peripheral CD34+ counts remain low after treatment with G-CSF alone, whether it was safe, and whether transplantation with the apheresis product was successful, as measured by time to engraftment of polymorphonuclear leukocytes (PMNs) and platelets (PLTs).

DETAILED DESCRIPTION:
A Phase 2, single-center, open-label study to assess the safety and hematological activity of plerixafor in patients with non-Hodgkin's lymphoma (NHL) or multiple myeloma (MM) who were predicted to be unable to mobilize ≥2*10^6 CD34+ cells/kg within 3 apheresis days. The only change to the standard of care was the addition of plerixafor to a G-CSF mobilization regimen on the day prior to apheresis.

Following screening procedures, eligible patients undergo mobilization with G-CSF (10 µg/kg every day) for 5 days and their peripheral blood (PB) CD34+ cell count was measured on the fifth day.

On Day 5, if the patient's peripheral CD34+ cell count was <5 cells/µl or ≥20 cells/µl, the patient did not enter this study and was treated as per the policy of the study site.

On Day 5, if the patient's peripheral CD34+ cell count was 5 to 7 cells/µl (inclusive), the patient did not undergo apheresis that day, but did receive plerixafor (240 µg/kg) that evening and G-CSF followed by apheresis the next morning. The evening dose of plerixafor followed the next morning by G-CSF and apheresis was repeated for up to a total of 3 days of apheresis or until ≥5*10^6 cells/kg are collected.

On Day 5, if the patient's peripheral CD34+ cell count was 8 to 19 cells/µl (inclusive), then he/she underwent apheresis that day. If this apheresis yield was <1.3*10^6 CD34+ cells/kg, then the patient was predicted to be unlikely to collect ≥2*10^6 CD34+ cells/kg in ≥3 days of apheresis and received plerixafor (240 µg/kg) that evening. However, if the apheresis yield on Day 5 was ≥1.3*10^6 CD34+ cells/kg, then the patient did not enter the study.

The next morning (Day 6), eligible patients received G-CSF (10 µg/kg) and began apheresis approximately 10 to 11 hours after the previous evening plerixafor dose. If the apheresis yield was at least double the apheresis yield on Day 5, then the patient received another 10:00 pm dose of plerixafor and underwent apheresis again the next morning (Day 7) after receiving G-CSF. The evening dose of plerixafor followed the next morning by G-CSF and apheresis was repeated for up to a total of 3 days of apheresis or until ≥5*10^6 cells/kg were collected.

All patients, after the completion of apheresis procedures (or after ≥5*10^6 cells/kg were collected), received high-dose chemotherapy in preparation for transplantation. Patients were transplanted with cells collected after receiving plerixafor with G-CSF. However, if there were insufficient cells, cells collected after receiving plerixafor with G-CSF could be pooled with cells collected after receiving G-CSF alone.

Hematological activity of plerixafor was evaluated by assessing the number of CD34+ cells harvested during apheresis.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria (Abbreviated List):

* Diagnosis of non-Hodgkin's lymphoma (NHL) or multiple myeloma (MM)
* Eligible for autologous transplantation
* <=3 prior regimens of chemotherapy (Rituxan is not considered chemotherapy for the purpose of this study)
* >4 weeks since last cycle of chemotherapy (Rituxan is not considered chemotherapy for the purpose of this study)
* Total dose of melphalan ≦200 mg
* Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell (WBC) count >3.0*10^9/L prior to first dose of G-CSF
* Absolute polymorphonuclear leukocyte (PMN) count >1.5*10^9/L prior to first dose of G-CSF
* Platelet (PLT) count >100*10^9/L prior to first dose of granulocyte colony-stimulating factor (G-CSF)
* Serum creatinine ≥2.2 mg/dL
* SGOT, SGPT and total bilirubin <2 times upper limit of normal (ULN)
* Negative for HIV
* CD34+ cell count between 5 and 19 CD34+ cells/ml after 5 days of mobilization with G-CSF alone

Exclusion Criteria (Abbreviated List):

* A co-morbid condition which, in the view of the investigator, renders the patient at high risk from treatment complications
* Failed previous stem cell collection or collection attempts
* A residual acute medical condition resulting from prior chemotherapy
* Active brain metastases or carcinomatous meningitis
* Active infection requiring antibiotic treatment
* Received prior radio-immunotherapy with Zevalin or Bexxar
* Received bone-seeking radionuclides (e.g., holmium)
* Received thalidomide, dexamethasone, and/or Velcade within 7 days prior to the first dose of G-CSF
* History of ventricular arrhythmias, including electrocardiogram (ECG)-documented premature ventricular contractions (PVCs), during the last 3 years
* Patients who previously received experimental therapy within 4 weeks of enrolling in this protocol or who are currently enrolled in another experimental protocol during the mobilization phase
* Had an apheresis yield >1.3*10^6 CD34+ cells/kg on Day 5 (Applicable only to patients who, after 5 days of G-CSF mobilization, have peripheral blood (PB) CD34+ count of 8-19 cells/µl inclusive).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-04; Primary Completion 2005-07 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Duke University Medical Center - Adult BMT Program, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began in April 2005 and the study was terminated in August 2006. Target enrollment was 15 patients, however the trial was terminated early after five patients were enrolled.
Groups:
- All Patients: Mobilization with Granulocyte Colony Stimulating Factor (G-CSF) (10 µg/kg once a day) for 5 days. Patients received once daily plerixafor treatment (240 mg/kg) in the evening (10 to 11 hours prior to apheresis) for up to 3 days if peripheral blood CD34+ cell counts on Day 5 met the entry criteria. Morning doses of G-CSF (10 µg/kg) continued throughout apheresis.
Period: Treatment Period
Arm/Group | All Patients
Started | 5
Completed | 4 (Failed mobilization due to <2 fold yield after one day of plerixafor treatment)
Not Completed | 1
Not completed — Failed Mobilization | 1
Period: Follow-up Period
Arm/Group | All Patients
Started | 5 (Participants who had transplants.)
Completed | 3
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5
Disease Diagnosis [Number; unit: participants] — One patient with HD was entered into the study even though there was no indication of MM or NHL (an inclusion criteria).
  participants
    Multiple Myeloma (MM) | 1
    Non-Hodgkin's lymphoma (NHL) | 3
    Hodgkin's disease (HD) | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved ≥2*10^6 CD34+ Cells/kg Following Treatment With Plerixafor 240 µg/kg and G-CSF for up to 3 Consecutive Days
Description: The number of patients with a circulating CD34+ count >= 5 and < 20 cells/ml after 5 days of mobilization with G-CSF alone who achieved cumulative apheresis yields of ≥2*10^6 CD34+ cells/kg within 3 days of apheresis after receiving G-CSF plus plerixafor. Outcome was based on laboratory results from a central lab.
Time Frame: approximately days 6-9
Population: All patients who received plerixafor.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 5
participants
  Participants with ≥2*10^6 CD34+ cells/kg | 3
  Participants with <2*10^6 CD34+ cells/kg | 2

2. Secondary Outcome: Overall Participants Counts of Adverse Events
Description: Numbers of participants with adverse events (AEs) collected from Day 1 (start of G-CSF Mobilization) to 12 months after transplantation. AEs were reported regardless of relationship to study treatment. The investigator graded each AE using the World Health Organization (WHO) Adverse Event Grading Scale and provided assessments of seriousness and relatedness to study treatment.
Time Frame: up to 13 months
Population: Safety Population defined as all participants who received G-CSF and/or plerixafor.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 5
participants
  Participants Reporting At Least One AE | 5
  Participants Reporting a Severe AE | 4
  Participants Reporting a Life-threatening AE | 2
  AE Relation to Drug: Not Related or Probably Not | 3
  AE Relation to Drug: Possibly Related | 2
  AE Relation to Drug: Probably or Definitely Relate | 0
  Serious Adverse Events | 4
  AEs Leading to Discontinuation | 0

3. Secondary Outcome: The Fold Increase in Peripheral Blood CD34+ Cells Following the First Dose of Plerixafor
Description: The fold increase was measured by fluorescence activated cell sorting (FACS) analysis and expressed as a ratio. Fold increase = pre-apheresis PB CD34+ cells/µL)/(pre-plerixafor dosing PB CD34+ cells/µL).
  This study was terminated early and analysis was not done.
Time Frame: Days 5-6
Population: This study was terminated early and analysis was not done.
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Days to Polymorphonuclear Leukocyte (PMN) Engraftment
Description: The median number of days to PMN engraftment criteria was PMN counts ≥ 0.5*10^9/L for 3 consecutive days or ≥ 1.0*10^9/L for 1 day. Time to engraftment corresponded to the first day that criteria were met.
  This study was terminated early and analysis was not done.
Time Frame: 2 months
Population: This study was terminated early and analysis was not done.
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Days to Platelet (PLT) Engraftment
Description: The median number of days to platelet (PLT) engraftment criteria was ≥ 20*10^9/L platelets without transfusion for the preceding 7 days. Time to engraftment corresponded to the first day that criteria were met.
  This study was terminated early and analysis was not done.
Time Frame: 2 months
Population: This study was terminated early and analysis was not done.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Graft Durability at 12 Months After Transplantation
Description: Participants with durable grafts. Graft durability was assessed by complete blood count (CBC) and differential analysis at 12 months post-transplantation.
  This study was terminated early and analysis was not done.
Time Frame: 13 months
Population: This study was terminated early and analysis was not done.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All treatment-emergent AEs are summarized. An event whose onset was on or after the first administration of study treatment (either G-CSF or plerixafor) was considered treatment-emergent.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Each AE table includes events regardless of reported relationship to study treatment or grade.
Groups:
- All Patients: All patients (3 NHL, 1 MM, and 1 HD).
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=5)
Acute myocardial infarction (Cardiac disorders) | 1 — Acute MI: Onset 15 days after last plerixafor dose, occurred during stem cell infusion, and assessed unrelated.
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=5)
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Infection (Infections and infestations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Limited enrollment due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.